CLINICAL TRIAL: NCT04922853
Title: Comparison of the Pathological Effect Between 2 and 4 Cycles Neoadjuvant CAPOX for Low/Intermediate Risk II/III Rectal Cancer：a Prospective, Non-inferior, Randomized, Controlled Trial
Brief Title: Comparison of the Pathological Effect Between 2 and 4 Cycles Neoadjuvant CAPOX for Low/Intermediate Risk II/III Rectal Cancer
Acronym: COPEC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: West China Hospital (Other)
Collaborators: The Third People's Hospital of Chengdu (Other); Chengdu Fifth People's Hospital (Other); Peking Union Medical College (Other); Peking University Cancer Hospital & Institute (Other); Sun Yat-sen University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Yunnan Cancer Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Sichuan Provincial People's Hospital (Other); Nanchong Central Hospital (Other Government); Dazhou Central Hospital (Other); Leshan People's Hospital (Unknown); GeneCast Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ziqiang Wang,MD, professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC-CT-2021
Record Dates: First submitted 2021-06-04; First posted 2021-06-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Rectal Cancer; Neoadjuvant Chemotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2 cycles group (Experimental): patients which recruited have 2 cycles Capox regimen (oxaliplatin: 130 mg/m2 iv d 1, capecitabine: 1000 mg/m2 bid d 1-14, repeated at 3 week intervals), then those patients with no sever chemotheraputic AE, have TME operation after reevaluation and randomization.
  Interventions: Drug: Capox chemotherapy
- 4 cycles group (Other): patients which recruited have 2 cycles Capox regimen (oxaliplatin: 130 mg/m2 iv d 1, capecitabine: 1000 mg/m2 bid d 1-14, repeated at 3 week intervals), then those patients with no sever chemotheraputic AE, have two more cycles chemotherapy and TME operation after reevaluation and randomization.
  Interventions: Drug: Capox chemotherapy

INTERVENTIONS:
Drug: Capox chemotherapy — oxaliplatin: 130 mg/m2 iv d 1, capecitabine: 1000 mg/m2 bid d 1-14, repeated at 3 week intervals

SUMMARY:
To compare the pathological effect between 2 cycles and 4 cycles of Capox regimen as neoadjuvant chemotherapy for low/ intermediate risk stage II/III rectal cancer.

DETAILED DESCRIPTION:
Neoadjuvant Chemotherapy alone has showed much benefit for low/ intermediate risk stage II/III rectal cancer which would be verified by the PROSPECT trial. However, the effect of the Neoadjuvant chemotherapy was heterogeneous in different patients. It's important to verify those chemo-resistant cases as early as possible. So that, this trial will compare the pathological effect between 2 cycles and 4 cycles of Capox regimen as neoadjuvant chemotherapy for low/ intermediate risk stage II/III rectal cancer to explore whether those chemotherapeutic non-responders after 2 cycles Capox was non-inferior to those after 4 cycles chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old; No gender limitation;
2. Patients diagnosed with low/intermediate risk stage II/III rectal cancer under MRI and transanal ultrasound,defined as: low:T3a-bN0-1M0, EMVI (±), MRF (-) (≥2mm); Middle-high rectal cancer: T3a-cN0-1M0, EMVI (±), MRF (-) (≥2mm); No more than 3 lymph nodes with short diameter over 8mm or highly suspected metastases; Patients with very low rectal cancer who met the above criteria and could achieve negative circumferential resection margin under ELAPE surgery could be included in the group
3. tumor located <=12cm from anal verge by colonoscopy or anal examination
4. no distant metastasis confirmed by CT examination;
5. rectal adenocarcinoma confirmed by pathology,
6. ECOG score: 0-1;
7. Patients with primary rectal cancer who did not receive surgery (except palliative stomy), radiotherapy, systemic chemotherapy or other anti-tumor therapy before enrollment;
8. Main organs function normally, that is, meet the following characteristics: ① Blood routine examination criteria should meet: Hb ≥9g/dL, WBC ≥ 3.5/4.0×109/L, neutrophils ≥ 1.5×109/L, PLT≥ 100×109/L. ② Biochemical tests should meet the following criteria: CREA and BIL ≤ 1.0 times upper limit of normal (ULN), ALT and AST≤ 2.5 times upper limit of normal (ULN), alkaline phosphatase (ALP) ≤2.5×UNL, total bilirubin (TBIL) ≤1.5×UNL.
9. No history of allergy to platinum drugs when no 5-FU drugs are allergic;
10. Women of childbearing age must have had a pregnancy test (serum or urine) 7 days prior to enrolment, be negative, and be willing to use an appropriate method of contraception during the trial and 8 weeks after the last dosing. For men, surgical sterilization or consent to use an appropriate method of contraception during the trial or for 8 weeks after the last dosing;
11. Subjects volunteered to participate in this study, signed the informed consent, and showed good compliance and followed up.

Exclusion Criteria:

1. patients suspect to Lynch syndrome;
2. Patients showed distant metastasis during treatment;
3. Previously or coexisting malignancies (including concurrent colon cancer), except for cured basal cell carcinoma of the skin and carcinoma in situ of the cervix;
4. pregnant or breastfeeding women;
5. Patients with severe cardiovascular diseases and diabetes that is not easily controlled;
6. People with mental disorders;
7. Severe infection;
8. sever renal disfunction;
9. History of gastrointestinal fistula, perforation, bleeding, or severe ulcer;
10. Allergic to 5-FU or platinum;
11. The presence of serious gastrointestinal diseases that affect the absorption of oral chemotherapeutic drugs; (12) Participants in additional clinical trials within 4 weeks prior to the start of treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Estimated)
Dates: Start 2021-08-26 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
pathological Tumor Regression Grade evaluation | 12 weeks
  pTRG

SECONDARY OUTCOMES:
rate of chemotherapeutic complication | 12 weeks
3-year overall survival | 3 year after recruiting
  the cumulative overall survival rate of the patients(events defined as all caused death)
disease free survival | 3 year after recruiting
  the cumulative disease free survival rate of the patients(events defined as tumor recurrence at any sites)
cumulative distant recurrence rate | 3 year after recruiting
  cumulative recurrence rate of Rectal cancer after the radical surgery outside the pelvic cavity
cumulative local recurrence rate | 3 year after recruiting
  cumulative recurrence rate of Rectal cancer after the radical surgery within the pelvic cavity or in the wounds

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Genecast Biotechnology Co., Ltd, Wuxi, Jiangsu
  - the Third People'S Hospital of Chengdu, Chengdu, Sichuan
  - West China Hospital, Chengdu, Sichuan
  - The Third Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shen Y, Shi W, Huang C, Gong X, Wei M, Meng W, Deng X, Wang Z; COPEC groups. Comparison of the pathological response to 2 or 4 cycles of neoadjuvant CAPOX in II/III rectal cancer patients with low/intermediate risks: study protocol for a prospective, non-inferior, randomized control trial (COPEC trial). Trials. 2023 Jun 13;24(1):397. doi: 10.1186/s13063-023-07405-x. PMID 37312165